CLINICAL TRIAL: NCT05312476
Title: Clinical Study of the Safety, Tolerability and Preliminary Efficacy of Chimeric Antigen Receptor T Cells (CAR-T) Targeting Igβ Targets in Patients With Igβ-positive Refractory Relapsed Non-Hodgkin's Lymphoma
Brief Title: Clinical Study on CAR-T Targeting Igβ Targets in Refractory Relapsed Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R/R B-NHL 02
Record Dates: First submitted 2022-03-21; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Relapsed/Refractory B-cell Non-Hodgkin's Lymphoma
Keywords: CAR-T Cells targeting Igβ targets; Relapsed Refractory B-cell Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Immunotherapy, Adoptive; Cell- and Tissue-Based Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chimeric Antigen Receptor T Cells (CAR-T) Targeting Igβ Targets (Experimental): Chimeric antigen receptor T cells targeting Igβ targets (CAR-T)
  Interventions: Drug: Chimeric Antigen Receptor T Cells (CAR-T) Targeting Igβ Targets

INTERVENTIONS:
Drug: Chimeric Antigen Receptor T Cells (CAR-T) Targeting Igβ Targets — 1. Dose escalation studies:3 dose groups in total: expect 3-6 cases in each group, and dose set at 1×106/kg，3×106/kg，6×106/kg.
  2. Dose extension study:3 cases (1 dose group).
  Other Names: Chimeric antigen receptor-modified T (CAR-T) cell therapy

SUMMARY:
Aim of this study will evaluate the safety, tolerability and preliminary efficacy of chimeric antigen receptor T cells (CAR-T) targeting Igβ targets in patients with Igβ-positive refractory relapsed non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
Non-Hodgkin's lymphoma is a group of malignant neoplasms of the lymphatic system originating from B or T cells, of which 60-70% of patients have B-cell-derived lymphoma (B-NHL). Although rituximab in combination with chemotherapy has significantly improved the prognosis of B-cell lymphoma, some patients still have primary resistance or relapse. In recent years, breakthroughs have been made in the treatment of B-cell tumors with Chimeric Antigen Receptor-Modified T Cells (CART), the investigators therefore constructed CAR-T cells targeting Igβ to investigate the safety and efficacy of CAR-T cells with this target for the treatment of r/r B-NHL.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signing of informed consent and good compliance.
2. Age ≥ 6 years.
3. Previously treated with 2 or more lines of therapy.
4. Has a measurable target lesion.
5. ECOG 0-1#.
6. Have appropriate organ function, subject to the following criteria (except for abnormal liver function due to tumor infiltration): AST≤3 times upper limit of normal#ALT≤3 times upper limit of normal# TB≤2 times ULN, unless combined with Gilbert's syndrome #Patients with Gilbert's syndrome with TB≤ 3 times ULN and DB≤ 1.5 times ULN can be include # Scr ≤1.5 times ULN or CCr≥60 ml/min# Lung function≤Level 1; dyspnea(CTCAE v5.0),and blood oxygen saturation without oxygen absorption> 91%# INR≤1.5 times ULN# aPTT≤1.5 times ULN.
7. negative blood/urine pregnancy test in women of childbearing age within 7 days prior to cell infusion, and any male and female patients of childbearing potential must agree to use an effective method of contraception throughout the study and for at least six months after the study treatment is administered.
8. Pass the T-cell amplification test.
9. Have adequate venous access to single or venous blood and no other contraindications to leukocyte isolation.
10. Estimated survival time ≥3 months.

Exclusion Criteria:

1. Prior malignancy (other than Relapsed Refractory B-cell Non-Hodgkin's Lymphoma), except for cured malignant tumors with no active lesions for 3 years; Adequate treatment of inactive lesions in non-melanoma skin cancer, malignant tonsilloma or carcinoma in situ.
2. Have used immunosuppressants or hormones within 2 weeks prior to signing informed consent, or plan to have to use immunosuppressants or high-dose hormones (e.g. prednisone >15mg) after signing informed consent, specifically systemic treatment, excluding treatment with topical or inhaled corticosteroids.
3. The presence of bacterial, fungal, viral, mycoplasma or other types of infection that, in the judgment of the investigator, are difficult to control.
4. HIV, Syphilis or COVID-19 infection.
5. Active hepatitis B or active hepatitis C.
6. Previous or current CNS disease other than this disease, such as seizures, cerebrovascular ischaemia/hemorrhage, dementia, cerebellar disease or any CNS-related autoimmune disease.
7. A history of cardiac angioplasty or stent placement within 12 months prior to signing the informed consent form, or a history of myocardial infarction, unstable angina or other clinically significant heart disease.
8. Patients with primary immunodeficiency.
9. Have had a severe tachyphylaxis to any of the drugs to be used in this study.
10. Live vaccination within 6 weeks prior to screening.
11. Pregnant or breasting-feeding women.
12. Active autoimmune diseases.
13. Active acute or chronic graft-versus-host disease (GVHD) at the time of signing the informed consent form.
14. Received an allogeneic hematopoietic stem cell transplant within 6 months prior to signing the informed consent form.
15. Participated in an investigational clinical trial of any other drug within 30 days prior to signing the informed consent form.
16. Conditions deemed by the researcher to be inappropriate for participation in this clinical trial.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2025-02-10 (Estimated); Study Completion 2025-02-10 (Estimated)

PRIMARY OUTCOMES:
DLT | Measured from start of treatment until 28 days after last dose
  DLT occurring within 28 days of the last dose.
Adverse events profile | Measured from start of treatment until 28 days after last dose
  Number of participants with adverse events. Frequencies of toxicities based on the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 5.0 will be tabulated.

SECONDARY OUTCOMES:
Objective Response Rate | up to 3 months
  Proportion of CR and PR subjects will be assessed at 3 months post-infusion.
Duration of Response | up to 12 months
  Duration of overall response will be assessed from the first chimeric antigen receptor T cells (CAR-T) targeting Igβ targets given to progression, death or last follow-up.
Progression-free survival | up to 12 months
  To measure the duration of response to chimeric antigen receptor T cells (CAR-T) targeting Igβ targets over a follow-up period of 12 months.
Overall Survival | up to 12 months
  OS will be assessed from the first chimeric antigen receptor T cells (CAR-T) targeting Igβ targets given to death or last follow-up.
Peak Plasma Concentration | Measured from start of treatment until 28 days after last dose
  the peak amplification of Igβ-CART in peripheral blood.
Time to Peak Amplification | Measured from start of treatment until 28 days after last dose
  the time to peak amplification of Igβ-CART in peripheral blood.
AUC0-28 | Measured from start of treatment until 28 days after last dose
  the area under the curve (AUC0-28) obtained by plotting the number of CAR-T cells in serum against the visit time from 0 to 28 days after reinfusion.
PD | Measured from start of treatment until 28 days after last dose
  Pharmacodynamics is the peripheral blood B-cell ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Depei Wu, M.D, Study Chair — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China